CLINICAL TRIAL: NCT05005871
Title: Comparison of the Effectiveness of Intramuscular and Transmucular Quadratus Lumborum Blocks Quality in Postoperative Pain
Brief Title: Comparison of Quadratus Lumborum Intramuscular and Transmuscular in Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, MD, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNUD-CTR-FK150621-001
Record Dates: First submitted 2021-06-15; First posted 2021-08-16 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative; Pain, Acute; Cesarean Section Complications
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum intramuscular block (Active Comparator): The quadratus lumborum intramuscular block will be performed immediately at the end of the surgery. Administration of 0.4 mL of 0.25% bupivacaine will be carried out under ultrasound guidance and performed by experienced anesthesiologists.
  Interventions: Other: Quadratus lumborum block after C-section surgery as postoperative pain management
- Quadratus lumborum transmucular block (Active Comparator): The quadratus lumborum transmuscular block will be performed immediately at the end of the surgery. Administration of 0.4 mL of 0.25% bupivacaine will be carried out under ultrasound guidance and performed by experienced anesthesiologists.
  Interventions: Other: Quadratus lumborum block after C-section surgery as postoperative pain management

INTERVENTIONS:
Other: Quadratus lumborum block after C-section surgery as postoperative pain management — To manage postoperative pain, the subjects will be allocated to either QLB or QLTB group to receive the respective intervention.

SUMMARY:
Acute pain is reported in approximately 80% of patients undergoing postoperative care for various types of surgical procedures in the United States. Another study reported patient postoperative pain intensity with 75% with severe pain in the first 1 to 2 postoperative days and 38% reporting moderate to severe pain at 14 postoperative days. Several modalities have been used as the standard for the management of pain postoperative C-sections.

One of the postoperative analgesic modalities for SC is quadratus lumborum block (QLB). This technique has advantages in relieving postoperative pain after C-section because it is considered to be able to relieve visceral pain as well as somatic pain. The transmuscular QLB (QLBT) approach is one of the most frequently used. This technique was found to be effective with regard to the distribution of analgesics to the paravertebral spaces which is the hallmark of QLB. However, this technique was found to be difficult to perform. Difficulties were reported related to the position of the procedure i.e. lateral or sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Underwent C-section with subarachnoid block
* Aged 18-35 years old.
* ASA preoperative physical status 1-2

Exclusion Criteria:

* Coagulopathy
* Anatomic abnormalities of the abdomen
* History of allergy to local anesthesia
* History of hyperalgesia
* History of drug abuse (sedatives, opioids, paracetamol, or other pain relievers)
* Require postoperative intensive care
* Refuse to participate in research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Up to 24 hours after surgery
  Postoperative pain intensity measured by Visual Analog Scale (VAS), 0=no pain, 100=worst pain
Postoperative morphine requirements | Up to 72 hours after surgery
  Total delivered morphine dose after surgery to alleviate postoperative pain (measured by total delivered dose recorded on the Patient-Controlled Analgesia tool)

CONTACTS AND LOCATIONS:
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided